CLINICAL TRIAL: NCT00198250
Title: Venlafaxine for Hot Flashes After Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Janet S. Carpenter, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0308-07; NINR/NIH R01 NR05261
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer survivorship; hot flashes; treatment
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: venlafaxine — Venlafaxine taper dose from 37.5mg for one week to 75 mg for 3 weeks
  Other Names: Effexor

SUMMARY:
The purpose of this study is to evaluate Venlafaxine as a treatment option for hot flashes in breast cancer survivors. The goals of this study are to assess the effectiveness and toxicity of venlafaxine hydrochloride and identify the psychological, behavioral, and physical outcomes associated with relief of hot flashes in women following treatment for breast cancer.

DETAILED DESCRIPTION:
Hot flashes are the most severe and fourth most prevalent menopausal symptom reported by women with breast cancer. Hot flashes affect over 65% of this population, with 59% rating the symptom as severe and 44% reporting they are extremely distressed by the symptom. Despite the high prevalence, severity and distress associated with this symptom, the scientific basis for managing hot flashes in women with breast cancer is limited. This randomized, double-blind, placebo-controlled crossover trial examines the effectiveness and toxicity of sustained release venlafaxine hydrochloride (37.5 mg po qd) on hot flashes in women following treatment for breast cancer. Venlafaxine is a phenylethylamine derivative that potently inhibits the reuptake of neuronal serotonin and norepinephrine and weakly inhibits the reuptake of dopamine. A secondary aim of this project is to examine the impact of hot flashes on psychological, behavioral, and physical outcomes. This study is based on the Wickham Symptom Management Model which depicts interrelationships between symptoms, symptom management strategies, and symptom management outcomes. Participants (n = 80) who are at least one month post-completion of surgery, radiation, and/or chemotherapy and who have been on tamoxifen (if prescribed) for at least six weeks will complete a two-week baseline hot flash assessment and be randomized to one arm of the crossover trial. At the end of the first six-week arm, participants will crossover to the opposite study arm for an additional six weeks. Outcomes to be assessed include effectiveness of the intervention (hot flash frequency, severity, distress and magnitude), toxicity of the intervention (subjective preference, side effects), psychological outcomes (mood disturbance), behavioral outcomes (quality of life, interference with daily activities) and physical outcomes (fatigue and sleep disturbance). Hot flashes will be measured daily, using a subjective, prospective diary methodology, and weekly, using objective state-of-the art 24-hour physiological monitoring of sternal skin conductance. Other outcomes will be measured weekly. Compliance with the intervention/placebo will be assessed weekly using medication blister pack cards. Timing of outcome assessments is based on limitations of the physiological monitoring device and expected timing of treatment effects. Summary statistics (i.e., mean, slope, maximum response, range, proportion, achievable difference) will be used to effectively reduce the design to a 2 X 2 crossover and data will be analyzed accordingly (i.e., t-tests, linear regression, GEE, mixed model). Study findings will significantly contribute to the scientific basis of hot flash management in women following treatment for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* women at least 21 years of age
* willing and able to provide informed consent
* first time diagnosis of breast cancer
* no other history of cancer
* considered disease free at time of study enrollment
* at least four weeks post-completion of surgery, radiation, and/or chemotherapy for non-metastatic cancer
* experiencing daily hot flashes
* desirous of treatment for hot flashes, but not concurrently using any other hot flash treatments
* living within 60 miles of Indianapolis
* able to read, write and speak English

Exclusion Criteria:

* current treatment with antidepressants for depression, neuropathic pain or hot flashes
* diagnosis of metastatic breast cancer (stage IV)
* treatment for hot flashes within the past four weeks, including (a) soy supplements; (b) botanicals, such as dong quai (Angelica sinensis), black cohosh, ginseng, gotu kola, licorice root, chaste tree, sage, or wild yam root; (c) vitamin E; or (d) prescription medications, such as clonidine hydrochloride or megestrol acetate.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2000-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Assess the effectiveness venlafaxine hydrochloride versus placebo in alleviating hot flash frequency, severity, distress, and magnitude in women following treatment for breast cancer. | completed

SECONDARY OUTCOMES:
Identify the psychological, behavioral, and physical outcomes associated with relief of hot flashes in women following treatment for breast cancer. | completed

CONTACTS AND LOCATIONS:
Overall Officials: Janet S Carpenter, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Carpenter JS, Storniolo AM, Johns S, Monahan PO, Azzouz F, Elam JL, Johnson CS, Shelton RC. Randomized, double-blind, placebo-controlled crossover trials of venlafaxine for hot flashes after breast cancer. Oncologist. 2007 Jan;12(1):124-35. doi: 10.1634/theoncologist.12-1-124. PMID 17227907